CLINICAL TRIAL: NCT07127146
Title: Role of Opioidergic and Noradrenergic Systems in Central Parkisonian Pain
Brief Title: Opioidergic and Noradrenergic Systems in Central Parkisonian Pain
Acronym: PAINPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_0721
Record Dates: First submitted 2025-06-18; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Pain; Parkinson's disease; Noradrenergic system; Opioidergic system; PET-MRI
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — carfentanil

STUDY DESIGN:
Intervention Model Description: Participants are assigned in 3 parallel groups without randomization :
  * group1 20 patients analyzable with Parkinson's disease suffering from central pain (PD-P)
  * Group 2 20 patients analyzable with Parkinson's disease without central pain (PD-NP) matched for sex and age.
  * Group 3 15 healthy volunteers analyzable (HC) matched for sex and age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD-P (Parkinson's patient with pain) (Experimental): Parkinson's patients suffering from chronic and central pain and with a VAS score of at least 4 points.
  They will perform 2 different PET MRI with radiotracer , one using [11C]Carfentanil and the other one using [11C]Yohimbine
  Interventions: Other: PET-MRI exam with administration of [11C]Carfentanil; Other: PET-MRI exam with administration of [11C]Yohimbine
- PD-NP (Parkinson's patient with no pain) (Experimental): Parkinson's patients without chronic and central pain and with a VASscore below 3 points They will perform 2 different PET MRI with radiotracer , one using [11C]Carfentanil and the other one using [11C]Yohimbine
  Interventions: Other: PET-MRI exam with administration of [11C]Carfentanil; Other: PET-MRI exam with administration of [11C]Yohimbine
- Healthy volunteers (Experimental): Healthy volunteers without chronic pain and with a VAS score below 3 points They will perform a PET MRI with the [11C]Carfentanil radiotracer
  Interventions: Other: PET-MRI exam with administration of [11C]Carfentanil

INTERVENTIONS:
Other: PET-MRI exam with administration of [11C]Carfentanil — Recording of functional neuroimaging data will begin immediately after intravenous injection of [11C]Carfentanil and will last for 51 minutes in a resting state. The dose will be 250 MBq/kg +-10 %.
Other: PET-MRI exam with administration of [11C]Yohimbine — Recording of functional neuroimaging data will begin immediately after intravenous injection of [11C]Yohimbine and will last for 70 minutes in a resting state. The dose will be 370 MBq/kg +- 10 %.
  Arms: PD-NP (Parkinson's patient with no pain); PD-P (Parkinson's patient with pain)

SUMMARY:
The goal of this study is to evaluate the differences in functional physiopathology of the opioid and noradrenergic systems between Parkinson's patients with central pain and Parkinson's patients without central pain. Using PET-MRI data, investigators aim to observe opioids receptors availability using [11C]Carfentanil (µ opioid receptor agonist) and altered α2-AR density with [11C]Yohimbine (adrenergic α2 receptor antagonist).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease based on MDS-UPDRS criteria (Group 1 and 2)
* Dopaminergic therapy stable with stable dose for at least 4 weeks prior to J0
* Affiliate to a social security or similar system
* Having given written consent to participate in the study, free and informed.
* Having chronic pain more than 3 month (Group 1)
* Without chronic pain (Groupe 2 and 3)
* Having central pain using specific algorithm (Marques et al., 2019)
* Having pain intensity at least 4 on VAS (Visual Analogue Scale) during the last month (Group 1)
* Having pain intensity lower than 3 on VAS (Visual Analogue Scale) during the last month (Group 2 and 3)

Exclusion Criteria:

* Having atypical Parkinson's disease (Group 1 and 2)
* Parkinson's disease with disabling dyskinesia and/or severe tremor (Group 1 and 2)
* Any contraindications to having a brain MRI or PET scan (e.g., pacemaker, metal foreign body, claustrophobia, deep brain stimulation or apomorphin pump unable to be turn off)
* History of head trauma with loss of consciousness lasting more than 30 minutes
* Not agreeing to be informed in the event of incidental discovery of an abnormality on MRI or during neuropsychological assessment
* Presence of cognitive dysfunction (defined as MoCA score < 24)
* Severe depression (BDI > 29)
* unable to stop the opioid treatment the week before the imaging exam ( e.g., Antarène codéine, Claradol codéine, Codoliprane, Dafalgan codéine, Euphon, Klipal, Lindilane, Néo-codion, Paderyl, Prontalgine, Pulmoserum, Tussipax ; Opium : Izalgi, Lamaline, Colchimax, Dropizal ; Morphine : Actiskenan, Moscontin, Oramorph, Sevredol, Skenan ; Buprénorphine : Bupensan, Buvidal, Orobupre, Sixmo, Suboxone, Subutex, Temgesic, Zubsolv ; Dihydrocodéine : Dicodin ; Hydromorphone : Sophidone ; Nalbuphine : Nalpain ; Fentanyl : Abstral, Actiq, Breakyl, Durogesic, Effentora, Instanyl, Matrifen, Pecfent, Recivit ; Méthadone : Methadone AP-HP, Zorvon ; Oxycodone : Oxsynia, Oxycontin, Oxynorm, Oxynormoro ; Tramadol : Biodalgic, Contramal, Ixprim, Monoalgic, Monocrixo, Orozamudol, Skudexum, Topalgic, Zaldiar, Zamudol, Zumalgic)
* unable to stop any treatment
* Treated with level 1 analgesics (NSAIDs, acetaminophen) or coanalgesics (antidepressants, antiepileptics) unless treatment has been stable for at least 4 weeks prior to the study and does not interfere with the noradrenergic system (list above).
* Presenting or having presented a dependence on any addictive substance according to DSM-IV-TR criteria, with the exception of tobacco.
* Having used recreational drugs interfering with the opioid and noradrenergic systems (cannabis, CBD, opiates, MDMA, ecstasy) in the last 3 months or chronic use
* Pregnant women, women in labor or nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* Under psychiatric care
* Admitted to a health or social institution for purposes other than research
* Under legal protection (guardianship, curatorship)
* Participant in another interventional study with an exclusion period still in progress at pre-inclusion
* Having exceeded the annual amount of compensation authorized for participation in research protocols

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference between non-displaceable binding potential of radiotracer in brain region involved in pain | At the time of PET-MRI scan at Day 75
  Differences between binding potential (BPND )of [11C]Carfentanil on the µ-opioid receptor and [11C]Yohimbine on α2-AR in PD-P and PD-NP patients

SECONDARY OUTCOMES:
Correlation between BPND of both tracer and pain intensity of parkinsonian patient | At the time of PET-MRI scan at Day 75
  Correlation between BPND measured with the [11C]Carfentanil and the[11C]Yohimbine and the pain intensity of all PD patient measured with clinical scores
Pain matrix area | At the time of PET-MRI scan at Day 75
  Compare the resting functional connectivity in the pain matrix area (insula, pre frontal cortex, thalamus) between groups of patients with and without pain.
ASL measure | At the time of PET-MRI scan at Day 75
  Observation of the blood flow modification through ASL measure in the brain pain areas between PD-P and PD-NP patients

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane THOBOIS, PHD, Study Director — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU de Clermont-Ferrand Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU de Toulouse - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided
It is not definied yet